CLINICAL TRIAL: NCT06171165
Title: Screening the Patient for Oral Intake: Applicability of the Yale Swallow Protocol in Patients Across Disease Categories
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401146RINE
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Oral Intake; Dysphagia; Swallow Difficulty
Keywords: Swallow; Dysphagia; Screening
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized Patients Across Disease Categories: We included the patients, namely, patients with head-and-neck cancer, stroke, and Parkinson's disease, as well as the elderly patients in acute care settings.
  Interventions: Diagnostic Test: Yale Swallow Protocol

INTERVENTIONS:
Diagnostic Test: Yale Swallow Protocol — All the participants will receive the two swallow screenings, i.e., Yale Swallow Protocol and Speech-language therapist, to classify the participants into either "try swallow" or "NPO" status.

SUMMARY:
With 98 swallow screening tools already developed, dysphagia remains under-screened and undiagnosed. Even for patients at high risk of oropharyngeal dysphagia (i.e., hospitalized aged, post-stroke, Parkinson's disease, head and neck cancer, or those had ≥ 48 hours of endotracheal intubation), swallow screening is not systematically performed. Nurses, as front-line providers, are bombarded with patients' dysphagia. We witnessed patients' subsequent poor outcomes, including delayed oral intake, dependence on the feeding tube, increased pneumonia, prolonged hospital length of stay, and increased in-hospital.

Despite many calls for nurses to perform bedside screens for timely management, there is a lack of census on what tools to use (98 available, many claimed to be valid) and whether nurses are capable of safely performing these screens, especially when facing across-disease patients. Without a screening tool that is used universally across different diseases to assess whether patients can safely engage in oral intake, clinical healthcare professionals will face significant challenges in conducting the screening. Meanwhile, we found the common, shared items, i.e., consciousness, voice/speech, coughing, oral motor movements, and water drinking tests or swallowing trials, are included in most swallow screening tools, suggesting these items are essential basics for oral intake safely.

Therefore, instead of creating a new screening tool, the aim of this study is to extract the common, shared items among existing swallowing screening tools and assemble them into a swallow screening protocol that can be administered by nursing staff for triage whether inpatient populations are at risk of unsafe for oral intake. After conducting a systematic review and assessing the quality, we found the Yale Swallow Protocol was identified as a high-quality swallowing screening tool and was used for screening the risk of aspiration across diverse outpatients who were referred for further swallow assessment. However, whether the Yale Swallow Protocol can be implemented in acute care settings to screen for "oral intake" requires further warranted for its applicability. Therefore, this study aims to test the applicability (i.e., accuracy, responsiveness, time-spending, and safety) of the Yale Swallow Protocol when used to screen for 'oral intake,' with speech therapists' evaluations serving as the reference standard for inpatients across various disease categories.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with any of the following conditions: (a) head-and-neck cancer, (b) stroke, (c) Parkinson's disease, (d) post-extubated, and (e) aged above 65 years.
* aged above 18 years.

Exclusion Criteria:

* Patients will be excluded if they are (a) feeding-tube dependent (gastrostomy tube, nasogastric tube), (b) nil per os (NPO), or (c) with airborne-transmitted diseases (e.g., open tuberculosis or SARS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the acute care setting diagnosed with various conditions
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
responsiveness | the time receiving the screenings
  floor effect or ceiling effect of Yale Swallow Protocol
time-spending to execute Yale Swallow Protocol | the time receiving the screenings
  the mean and standard deviation
safety | the time receiving the screenings
  whether any unanticipated adverse effect exists when executing Yale Swallow Protocol

SECONDARY OUTCOMES:
responsiveness | the time receiving the screenings
  difficulty of Yale Swallow Protocol analyzed by Item Response Theory
parsimony | the time receiving the screenings
  shorten the Yale Swallow Protocol by Item Response Theory

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chia-Hui Chen, DNSc, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University School of Nursing, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang YC, Wu MS, Siao SF, Wang MJ, Xu YJ, Chen CC. Identifying High-Quality Non-Instrumental Dysphagia Screening Tools for Detection of Adult Dysphagia Case in Acute-Care Settings: A Systematic Review. Clin Otolaryngol. 2024 Nov;49(6):687-698. doi: 10.1111/coa.14194. Epub 2024 Jun 28. PMID 38940226